CLINICAL TRIAL: NCT01442428
Title: Randomized Controlled Trial for Corticosteroids Versus NSAIDs With or Without Adjunctive Atorvastatin for the Treatment for Paradoxical Tuberculosis Immune Reconstitution Inflammatory Syndrome
Brief Title: Paradoxical Tuberculosis Immune Reconstitution Inflammatory Syndrome (TB-IRIS) Treatment Trial
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: 2011 Thailand flooding led to loss of GMP pharmacy, project delays, and further regulatory challenges.
Sponsor: University of Minnesota (Other)
Collaborators: Pfizer (Industry); Minnesota Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WS967180
Record Dates: First submitted 2011-08-30; First posted 2011-09-28 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Immune Reconstitution Inflammatory Syndrome; Immune Reconstitution Syndrome; Tuberculosis; HIV-infection/Aids
Keywords: TB; AIDS; HIV; IRIS; immune reconstitution inflammatory syndrome; anti-inflammatory; treatment
MeSH Terms: conditions — Immune Reconstitution Inflammatory Syndrome; Tuberculosis; Acquired Immunodeficiency Syndrome | interventions — Dexamethasone; Calcium Dobesilate; Atorvastatin; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Steroid+Statin (Experimental): 1. Dexamethasone: 4 mg 3x daily for 2 weeks, then 2x daily for 1 week, then once daily for 1 week;
  2. Atorvastatin: 80 mg once daily (equivalent to 30mg ± 10mg with rifamycin co-administration)
  Interventions: Drug: Dexamethasone; Drug: Atorvastatin
- NSAID+Statin (Active Comparator): 1. Naproxen: 250 mg 3x daily for 2 weeks, then 2x daily for 1 week, then once daily for 1 week;
  2. Atorvastatin: 80 mg once daily (equivalent to 30mg ± 10mg with rifamycin co-administration)
  Interventions: Drug: Atorvastatin; Drug: Naproxen
- Steroid+Placebo (Active Comparator): 1. Dexamethasone: 4 mg 3x daily for 2 weeks, then 2x daily for 1 week, then once daily for 1 week;
  2. Placebo
  Interventions: Drug: Dexamethasone; Drug: Placebo
- NSAID+Placebo (Active Comparator): 1. Naproxen: 250 mg 3x daily for 2 weeks, then 2x daily for 1 week, then once daily for 1 week;
  2. Placebo
  Interventions: Drug: Naproxen; Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone: 4 mg 3x daily for 2 weeks, then 2x daily for 1 week, then once daily for 1 week
  Other Names: decadron
  Arms: Steroid+Placebo; Steroid+Statin
Drug: Atorvastatin — Atorvastatin: 80 mg once daily (equivalent to 30mg ± 10mg with rifamycin co-administration in this TB population)
  Other Names: Lipitor
  Arms: NSAID+Statin; Steroid+Statin
Drug: Naproxen — Naproxen: 250 mg 3x daily for 2 weeks, then 2x daily for 1 week, then once daily for 1 week
  Other Names: naproxen sodium; Aleve; Anaprox; Antalgin; Feminax Ultra; Flanax; Inza; Midol Extended Relief; Nalgesin; Naposin; Naprelan; Naprogesic; Naprosyn; Narocin; Proxen; Synflex; Xenobid
  Arms: NSAID+Placebo; NSAID+Statin
Drug: Placebo — Atorvastatin placebo
  Arms: NSAID+Placebo; Steroid+Placebo

SUMMARY:
Tuberculosis is the most common opportunistic infection (OI) in HIV-infected persons worldwide, including in South East Asia. Significant numbers of patients experience tuberculosis-related paradoxical immune reconstitution inflammatory syndrome (TB-IRIS) after ART initiation, yet the optimal treatment of TB-IRIS is unknown. A recent randomized-controlled trial showed the benefit of prednisone over placebo in reduction of days of hospitalization and invasive procedures. The investigators hypothesize that nonsteroidal anti-inflammatory drugs (NSAIDs) are as effective as corticosteroids for treatment of non-life threatening TB-IRIS in HIV-infected patients and hypothesize that adjunctive treatment with 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase inhibitors (Statins) may improve the outcomes. This is a randomized controlled trial with a 2x2 factorial design to test the relative benefit of corticosteroids, NSAIDS, and Statins for the symptomatic and immunologic control of TB-IRIS.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection documented by any locally licensed ELISA or rapid HIV test kit.
* Age >18 years
* Paradoxical TB-IRIS diagnosed by case definition (see section 5.2)
* Ability and willingness of the participant or legal guardian/representative to give informed consent. Receiving appropriate ART and anti-TB therapy, as judged by the site investigator

Exclusion Criteria:

* Inability to take oral medication;
* Receiving chemotherapy, immunosuppressant, corticosteroid, NSAID, or statin medications; (ASA is acceptable)
* Cannot or unlikely to attend regular clinic visits;
* Known allergy to NSAIDs, statins or corticosteroids;
* Liver transaminase > 2 times the upper limit of normal within 60 days of enrollment;
* History of myositis/myopathy;
* High Investigator Suspicion of anti-TB treatment failure due to TB-resistance or medication non-adherence;
* Receiving ongoing azole anti-fungal for treatment or secondary prophylaxis of cryptococcosis, histoplasmosis or penicilliosis;
* Serious co-morbidities, co-infections, or laboratory values who should not receive NSAIDs, steroid or statins, as judged by the site investigator;
* Minimal IRIS reaction which is unlikely to require treatment, as judged by the site investigator;
* Pregnancy (a negative urine pregnancy test at screening is required for women of childbearing potential) or breast feeding;
* Receiving a HIV treatment regimen containing a protease inhibitor at study entry.

Exclusion for Randomization A Only

* Life threatening TB-IRIS, as defined by:
* Acute respiratory failure; PaO2 < 60 on room air or;
* Altered mental status or;
* New focal neurological deficit or;
* Compression of the vital organs.
* Persons with uncontrolled diabetes mellitus;
* Impair kidney function, glomerular filtration rate <60 ml/min; within 72 hours of consent
* Uncontrolled congestive heart failure
* History of bleeding disorder;
* Platelet count <100,000/µL;
* History of significant gastrointestinal bleeding or ulceration;
* Prior adjunctive corticosteroid therapy for this TB episode for > 48 hr;
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Symptom Score at Day 7, as measured by the 10-point visual analog scale to quantify symptom severity. | Day 7
Change in serum C-reactive protein at Day 7 | Day 7

SECONDARY OUTCOMES:
Days of hospitalization combined with outpatient therapeutic procedures | 56 days
Study medicine discontinuation | 28 days
  (e.g. switching to open-label medication)
Karnofsky Performance Status Scale at day 7 and 28; | Day 7 and Day 28
Incidence of Adverse Events | 56 days
  DAIDS Grading Scale 3-5 events
Radiologic improvement at 2 weeks; | 14 days
Mortality | 56 days
CD4 count change | 28 days
Recurrence of IRIS manifestations within the 8 week study period | 56 days
ART or TB therapy discontinuation | 56 days
Incidence of sputum acid fast bacilli (AFB) smear positivity at day 28 | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Sasisopin Kiertiburanakul, MD, MHS, Principal Investigator — Mahidol University; David R Boulware, MD, MPH, Study Chair — University of Minnesota; Ubonvan Jongwutiwes, MD, Study Director — Memorial Sloan Kettering Cancer Center
Locations (3):
- Thailand (3):
  - Ramathibodi Hospital, Bangkok
  - Chiang Mai University, Chiang Mai
  - Bamrasnaradura Infectious Diseases Institute, Nonthaburi